CLINICAL TRIAL: NCT02292121
Title: Intestinal Permeability in Obesity of Intercellular Tight Junctions to Metabolic Complications
Brief Title: Intestinal Permeability in Obesity
Acronym: LEAKY GUT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of surgical controls
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institute of Cardiometabolism and Nutrition, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: P130402
Record Dates: First submitted 2014-11-12; First posted 2014-11-17 (Estimated); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Obesity; Metabolic Diseases; Nutrition Disorders; Body Weight
Keywords: Obesity; Intestinal permeability; Adipose tissue inflammation; Low grade systemic inflammation; Bariatric surgery
MeSH Terms: conditions — Obesity; Metabolic Diseases; Nutrition Disorders; Body Weight | interventions — Intestinal Barrier Function; lactitol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- obese group (Experimental): 40 obese subjects undergoing gastric bypass explored at baseline and 30 explored post-surgery at 6 months
  Interventions: Procedure: Intestinal permeability; Other: a solution of mannitol and lactitol
- non-obese control group (T1) (Active Comparator): 30 non-obese control subjects investigated for bio-clinical measures, IPT, zonulin, and LPS
  Interventions: Procedure: Intestinal permeability; Other: a solution of mannitol and lactitol
- non obese control group undergoing a surgery (T2) (No Intervention): 40 non-obese candidates to a surgery that gives access to surgical jejunal samples to measure the expression of tight junctions proteins

INTERVENTIONS:
Procedure: Intestinal permeability — 5h-intestinal permeability test 10-hour overnight fasting subject who first emptied his bladder drinks a solution of mannitol and lactitol. 2 hours after, the subject drinks 500mL of water in less than 30 minutes. All urine samples are collected during the 5h-test for measurement of lactitol and mannitol.
  Arms: non-obese control group (T1); obese group
Other: a solution of mannitol and lactitol
  Arms: non-obese control group (T1); obese group

SUMMARY:
In rodents, obesity is associated with changes in tight junctions' structure in small intestine, which impacts intestinal permeability and results in metabolic complications. Few data exist in human. We hypothesized that intestinal permeability is altered in obese subjects in comparison to lean subjects, linked to metabolic and inflammatory status and that these alterations are modified after gastric bypass.

DETAILED DESCRIPTION:
The regulation of the permeability of the intestinal barrier is essential in the molecular traffic between the lumen and the internal environment. It affects the absorption of nutrients and tolerance or immunization against foodborne non-self antigens that penetrate the barrier. In rodents, increased endotoxemia has been proposed as an important player in low-grade inflammation accompanying the development of obesity and metabolic disorders. In humans, the intestinal barrier function is altered in inflammatory bowel diseases (IBD, Crohn's disease, ulcerative colitis and celiac disease). The term "leaky gut" is used to describe a porous intestine with hyper-permeability associated with acute or chronic inflammatory diseases such as "systemic inflammatory response syndrome (SIRS),"acute inflammatory bowel disease (IBD for "inflammatory bowel disease").

Deficiencies of the barrier are also observed in extra-intestinal diseases (type-1 diabetes, food allergies, and autoimmune diseases). Impairments in tight junctions may precede clinical signs and constitute a risk factor for developing diseases or secondarily be altered and cause an increased entry of undesirable bacterial or nutritional antigens. The state of the intercellular tight junctions of the intestine controls the diffusion of molecules between cells. A deficiency of the intestinal barrier function is often associated with structural changes in the tight junctions resulting from loss of localization of protein or expression of genes and / or cellular signals such as ZO-1, occludin or tricellulin.

There are few studies about the condition of the intestinal barrier in the context of human obesity.

The objectives of our study are to :

* compare intestinal permeability in obese subjects with non obese subjects and after gastric bypass.
* search links between intestinal permeability and 1) metabolic and inflammatory bioclinical parameters 2) dietary profiles 3) microbiota

ELIGIBILITY:
Inclusion criteria :

- Control subjects T1:

1. Registered for social security
2. Signed consent form
3. male or female subject between 18 and 65 years old
4. Fasting plasma triglycerides < 1.5 g/l (< 1.7 mmol/l)
5. Fasting plasma total cholesterol < 2.5 g/l (< 6 mmol/l)
6. fasting glycaemia < 5,5 mmol/l
7. BMI <25kg/m² & >18 kg/m²
8. Mean systolic blood pressure <140 mmHg and mean diastolic blood pressure < 90 mmHg.

Control subjects T2

1. Registered for social security
2. Signed consent form
3. male or female subject between 18 and 70 years old
4. IMC<25kg/m² et >18 kg/m²
5. candidate to surgery giving access to jejunal samples

Obese subjects OB:

1. Registered for social security
2. Signed consent form
3. male or female subject between 18 and 65 years old
4. Candidate to bariatric surgery (bypass) with massive (IBMI >= 40 kg/m²) or severe obesity (BMI between 35 & 40 kg/m²) with at least one obesity-related comorbidity and with a stable weight (+/-5kg) for the last 3 months, after approval by a multidisciplinary team

Exclusion criteria :

- Control subjects T1:

1. Subject with a history of vascular symptomatic disease in the last 6 months before selection.
2. Subject receiving a treatment that can affect measured parameters
3. Pregnancy
4. Subject with acute or chronic disease that can affect measured parameters or to life-threatening. Including but not limited :

   1. Diabetic subjects
   2. Subject with kidney disease: nephrotic syndrome, chronic renal failure
   3. Subject having a gastrointestinal disorder or disease limiting intestinal absorption (celiac disease), bariatric surgery.
   4. Active inflammatory disease or a history of IBD
5. Subject in a situation that, according to the investigator's opinion could interfere with an optimal participation to the study or constitute a particular risk to the subject
6. Subject in an exclusion period after participating in another clinical trial
7. Adult person subject to legal protection or unable to consent.
8. Persons deprived of their liberty by judicial or administrative decision

Control subjects T2

1. Subject with a history of symptomatic vascular disease (myocardial infarction, angina syndrome threat, surgical or endovascular surgery, stroke, lower limb arteritis symptomatic) of less than 6 months
2. Subject with any acute or chronic disease which may influence the results of the study or to life-threatening. Including but not limiting:

   1. diabetic patients
   2. Subject with kidney disease: nephrotic syndrome, chronic renal failure and / or serum creatinine> 1.7 times the upper limit of the reference value
3. Adult person subject to legal protection or unable to consent.
4. Persons deprived of their liberty by judicial or administrative decision

Obese subjects candidates for surgery:

1. Subject receiving treatment systemically or topically, which may interfere with the evaluation of the parameters studied (NSAIDs, antibiotics in the previous month)
2. Any disease or psychosocial context making prolonged regular monitoring impossible, which also represents a contraindication for bariatric surgery.
3. Adult person subject to legal protection or unable to consent.
4. Persons deprived of their liberty by judicial or administrative decision

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-02-24 (Actual); Primary Completion 2016-03-17 (Actual); Study Completion 2016-03-17 (Actual)

PRIMARY OUTCOMES:
urinary lactitol / mannitol ratio by an intestinal permeability test (IPT) | before gastric bypass and 6 months after
  Measures of urinary lactitol / mannitol ratio by an intestinal permeability test (IPT) in obese patients before gastric bypass and 6 months after

SECONDARY OUTCOMES:
fasting zonulin serum concentrations | before gastric bypass and 6 months after
  Measures of fasting zonulin serum concentrations in obese patients before gastric bypass and 6 months after
LPS serum concentrations | before gastric bypass and 6 months after
  Measures of LPS serum concentrations in obese patients before gastric bypass and 6 months after
urinary lactitol / mannitol ratio by an intestinal permeability test (IPT) | inclusion and after one month
  Measures of urinary lactitol / mannitol ratio by an intestinal permeability test (IPT) in non-obese control subjects, performed twice with a one-month interval.
surgical samples during surgery (sub-cutaneous and visceral adipose tissue) | intraoperative

CONTACTS AND LOCATIONS:
Overall Officials: Christine POITOU, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Groupe Hospitalier Pitié-Salpêtrière, Paris, France